CLINICAL TRIAL: NCT00549796
Title: Randomized Comparison Angioplasty Outcomes at Hospitals With and Without On-site Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other); Maryland Medical Research Institute (Other)
Responsible Party: Principal Investigator, Thomas Aversano, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_000230; C-PORT E Trial
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Arteriosclerosis; Angina Pectoris
Keywords: coronary artery disease; angioplasty; stent; percutaneous coronary intervention; on-site cardiac surgery; randomized trial
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): PCI performed at a hospital with co-located (on-site) cardiac surgery
  Interventions: Other: Percutaneous coronary intervention (PCI)
- 2 (Other): PCI performed at a hospitals without co-located (on-site) cardiac surgery
  Interventions: Other: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Other: Percutaneous coronary intervention (PCI) — Patients undergo routine, clinically indicated PCI

SUMMARY:
Angioplasty is a procedure which opens blocked heart arteries using balloons and/or stents. Most U.S. states and all national heart organizations require that angioplasty be done only at hospitals that can also perform open heart surgery. The reason for this is that there is a risk that angioplasty can cause injury to the heart artery that might require open heart surgery to fix. Open heart surgery is a backup in case it is needed. The risk that open heart surgery will be needed is very small. Nevertheless, without more research, many state Departments of Health and all national heart organizations do not want to change the requirement for having on-site open heart surgery wherever angioplasty is performed. Some States already allow this; and European heart organizations already allow it, as well.

This study is designed to determine whether the safety and benefits of angioplasty are the same at hospitals that perform angioplasty either with or without open heart surgery backup.

Patient who enter the study have a heart catheterization at a hospital without a heart surgery program. If they need angioplasty, then they are randomized to either stay at the hospital without heart surgery for their angioplasty or to be transferred for the procedure to a hospital with heart surgery. For every four patients, three stay at the hospital without heart surgery and one is transferred.

The study is designed to show that there is no detectable difference between the safety and benefits of the procedure at the two types of hospital (with and without heart surgery). The cost of the procedure at the two hospital types is also compared.

ELIGIBILITY:
Inclusion Criteria:

Pre-catheterization:

* Must be undergoing diagnostic cardiac catheterization for suspected CAD
* Be at least 18 years of age
* Must not be pregnant (negative pregnancy test) or must not be of childbearing potential must be able to give informed consent.

Post-catheterization:

* Coronary artery disease judged to be clinically and angiographically significant
* Ability to perform PCI with equipment available at the local site
* Procedure risk judged to be not high (see below)

Exclusion Criteria:

Pre-catheterization:

* Inability to give informed consent
* ST-segment elevation myocardial infarction
* Pregnancy

Post-catheterization:

* High likelihood of requiring a device not available at the hospitals without SOS
* No need for PCI
* Need for coronary artery bypass surgery
* High procedural risk (see below)

High procedural risk criteria are:

* PCI of unprotected left main coronary artery
* PCI of left circulation lesion in the presence of critical (>70%) unprotected left main coronary artery lesion
* Poor left ventricular function (EF< 20%) and need to perform PCI in a vessel supplying significant myocardium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18876 (Actual)
Dates: Start 2006-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 weeks
MACE = death + MI + TVR | 9 Months

SECONDARY OUTCOMES:
emergency CABG | hosp DC, 6 wks, 3, 6 and 9 months
myocardial infarction | hosp DC, 6 wks, 3, 6 and 9 months
target vessel revascularization (TVR) | hosp DC, 6 wks, 3, 6 and 9 months
any subsequent revascularization (ASR) | hosp DC, 6 wks, 3, 6 and 9 months
heart failure and class | hosp DC, 6 wks, 3, 6 and 9 months
angina and class | hosp DC, 6 wks, 3, 6 and 9 months
stroke | hosp DC, 6 wks, 3, 6 and 9 months
composite adverse endpoint (MACE) | hosp DC, 6 wks, 3, 6 and 9 months
MACE = death + MI + TVR | hosp DC, 6 wks, 3, 6 and 9 months
MACE = death + MI + ASR | hosp DC, 6 wks, 3, 6 and 9 months
angiographic (end-procedure) complications (embolization, dissection, no reflow, etc) | hosp DC, 6 wks, 3, 6 and 9 months
angiographic (procedural) success (<20% residual stenosis and TIMI 3 flow) | hosp DC, 6 wks, 3, 6 and 9 months
completeness of revascularization | hosp DC, 6 wks, 3, 6 and 9 months
percent of patients with complete or partial revascularization | hosp DC, 6 wks, 3, 6 and 9 months
bleeding (non-CABG transfusion, vascular repair) | hosp DC, 6 wks, 3, 6 and 9 months
length of stay | hosp DC, 6 wks, 3, 6 and 9 months
total direct medical cost | hosp DC, 6 wks, 3, 6 and 9 months
major resource consumption patterns (hospital and ICU days, surgeries, hospitalizations) | hosp DC, 6 wks, 3, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aversano, MD, Study Director — Johns Hopkins University
Locations (60):
- United States (60):
  - Crestwood Medical Center, Huntsville, Alabama
  - Wellstar Cobb Hospital, Austell, Georgia
  - Southeast Georgia Health System, Brunswick, Georgia
  - Tanner Medical Center, Carrollton, Georgia
  - Hamilton Medical Center, Dalton, Georgia
  - Fairview Park Hospital, Dublin, Georgia
  - Spalding Regional Medical Center, Griffin, Georgia
  - West Georgia Health, La Grange, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Archbold Memorial Hospital, Thomasville, Georgia
  - Tift Regional Medical Center, Tifton, Georgia
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - Southern Maryland Hospital Center, Clinton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Bayonne Medical Center, Bayonne, New Jersey
  - Clara Maas Medical Center, Belleville, New Jersey
  - JFK Medical Center, Edison, New Jersey
  - Trinitas Hospital, Elizabeth, New Jersey
  - Robert Wood Johnson Medical Center, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua-West Jersey Hospital Marlton, Marlton, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Muhlenberg Regional Medical Center, South Plainfield, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Community Health and Wellness Center, Bryan, Ohio
  - University Hospitals Case Medical Center / Geauga Medical Center, Chardon, Ohio
  - University Hospital East Ohio State University Medical Center, Columbus, Ohio
  - Southview Medical Center, Dayton, Ohio
  - Fort Hamilton Hospital, Hamilton, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mt. Carmel St. Ann's Hospital, Westerville, Ohio
  - Legacy Meridian Park Hospital, Portland, Oregon
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Evangelical Community Hospital, Lewisburg, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - West Chester Hospital, West Chester, Pennsylvania
  - Memorial Hospital, York, Pennsylvania
  - Kingwood Medical Center, Kingwood, Texas
  - Mainland Medical Center, Texas City, Texas

REFERENCES:
- [Derived] Hiremath PG, Aversano T, Spertus JA, Lemmon CC, Naiman DQ, Czarny MJ. Sex Differences in Health Status and Clinical Outcomes After Nonprimary Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2022 Feb;15(2):e011308. doi: 10.1161/CIRCINTERVENTIONS.121.011308. Epub 2022 Jan 23. PMID 35067071
- [Derived] Aversano T, Lemmon CC, Liu L; Atlantic CPORT Investigators. Outcomes of PCI at hospitals with or without on-site cardiac surgery. N Engl J Med. 2012 May 10;366(19):1792-802. doi: 10.1056/NEJMoa1114540. Epub 2012 Mar 25. PMID 22443460